CLINICAL TRIAL: NCT06305143
Title: The Efficacy and Safety of Conbercept for Diabetic Macular Edema Combined With Severe Non-proliferative Diabetic Retinopathy: 12-month Results From a Prospective Multicenter Open Label Study
Brief Title: Efficacy and Safety of Conbercept for Diabetic Macular Edema Combined With Severe Non-proliferative Diabetic Retinopathy
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Shanghai Eye Disease Prevention and Treatment Center (Other)
Collaborators: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YFZXYDK202402
Record Dates: First submitted 2024-03-04; First posted 2024-03-12 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Diabetic Macular Edema
MeSH Terms: interventions — KH902 fusion protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- intravitreal Conbercept (Experimental): Participants with diabetic macular edema (DME) combined with severe non-proliferative diabetes retinopathy (sNPDR) were assigned to anti-VEGF therapy over 12 months.
  Interventions: Drug: Conbercept

INTERVENTIONS:
Drug: Conbercept — participants with diabetic macular edema (DME) combined with severe non-proliferative diabetes retinopathy (sNPDR) were assigned to anti-VEGF therapy over 12 months.

SUMMARY:
The goal of this prospective multicenter open label study is to evaluate the efficacy and safety of intravitreal injection Conbercept (IVC) for the treatment of diabetic macular edema (DME) combined with severe nonproliferative diabetes retinopathy (sNPDR).

The main questions it aims to answer are:

* mean changes in best corrected visual acuity (BCVA) and central macular thickness (CMT) in comparison with baseline at 12 months after initial treatment
* proportion of eyes with visual gain ≥15 letters in Early Treatment Diabetic Retinopathy Study (ETDRS) chart and ≥2-step improvement in Diabetic Retinopathy Severity Scale (DRSS) score after 12 months of the treatment
* proportion of eyes actually underwent PRP treatment after 3 and 12 months of the treatment
* mean changes in BCVA and CMT from baseline to monthly follow-up time point
* complications and adverse effects

ELIGIBILITY:
Inclusion Criteria:

* symptomatic patients aged 18 years or above with center involved diabetic macular edema in the involved eye and without clinically significant diabetic macular edema in the fellow eye defined on the basis of spectral-domain optical coherence tomography (OCT)
* central macular thickness (CMT) ≥300 μm measured by OCT
* the involved eyes diagnosed as severe non-proliferative diabetic retinopathy (sNPDR) confirmed by two independent experienced ophthalmologists based on the ETDRS standard seven field color fundus photographs

Exclusion Criteria:

* concomitant or previous macular diseases that may hinder visual improvement other than diabetic retinopathy (e.g., retinal vein occlusion, age-associated macular degeneration, uveitis, vitreomacular traction or epiretinal membrane)
* history of glaucoma or optic neuropathy of any kind
* previous vitreoretinal surgery or pan-retinal photocoagulation
* intravitreal injection anti-VEGF drugs within 6 months or intravitreal injection glucocorticoid within 3 months
* macular focal/grid laser photocoagulation within 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
improvement of visual acuity | from baseline to 12 months after initial intravitreal Conbercept injection
  mean change in best corrected visual acuity letter score

CONTACTS AND LOCATIONS:
Overall Officials: Tao Sun, Study Chair — Shanghai Eye Diseases Prevention & Treatment Center
Locations (1):
- Shanghai Eye Diseases Prevention &Treatment Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No